CLINICAL TRIAL: NCT00052572
Title: A Multicenter Phase II Study Of BMS 247550 (Epothilone B Analogue) In Indolent Lymphoproliferative Disorders
Brief Title: Ixabepilone in Treating Patients With Relapsed or Refractory Lymphoproliferative Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258542; MSKCC-02046; NCI-5342
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2006-04

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; Waldenström macroglobulinemia; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent mantle cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — ixabepilone

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ixabepilone in treating patients who have relapsed or refractory lymphoproliferative disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the frequency and duration of complete and partial response rates for patients with relapsed or refractory indolent lymphoproliferative disorders treated with ixabepilone.

Secondary

* Determine the time to progression and overall survival of patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive ixabepilone IV over 1 hour weekly for 3 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study within 1-1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed relapsed/recurrent or refractory indolent lymphoproliferative disorder of 1 of the following types:

  * Chronic lymphocytic leukemia

    * Absolute lymphocytosis greater than 5,000/mm^3
    * B-cell phenotype (CD 19, 20, or 23 positive) with more than 30% bone marrow lymphocytes
  * B-cell small lymphocytic lymphoma
  * Marginal zone B-cell lymphoma
  * Grade I-III follicle center cell lymphoma
  * Waldenstrom's macroglobulinemia
  * Mantle cell lymphoma
* At least 1 unidimensionally measurable lesion for patients with non-Hodgkin's lymphoma

  * At least 2 cm by conventional techniques
* No active brain metastases

  * Treated CNS disease allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3 (500/mm^3 if there is lymphomatous involvement of the bone marrow)
* Platelet count ≥ 50,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 2.5 times ULN (4 times ULN if there is liver involvement)

Renal

* Creatinine ≤ 2 times ULN OR
* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* No history of orthostatic hypotension
* No myocardial infarction, cerebrovascular accident, or transient ischemic attack within the past 3 months
* No New York Heart Association class III or IV congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension requiring manipulation of antihypertensive medications
* No evidence of any of the following by echocardiogram:

  * Acute ischemia
  * Significant conduction abnormality

    * Bifascicular block
    * 2^nd- or 3^rd-degree atrioventricular block

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other immunodeficiency
* No known severe hypersensitivity reaction to agents containing Cremophor EL
* No ongoing or active infection
* Febrile episodes up to 38.5° Celsius allowed in the absence of infection
* No other concurrent uncontrolled illness that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* No preexisting grade II or greater sensory neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior monoclonal antibodies (unless there is clearly documented evidence of disease progression after therapy)
* At least 3 months since prior radioimmunotherapy
* No prior allogeneic bone marrow transplantation

Chemotherapy

* At least 4 weeks since prior cytotoxic chemotherapy (6 weeks for mitomycin, nitrosoureas, or carmustine) and recovered
* No more than 4 prior chemotherapy regimens (including high-dose chemotherapy [HDC] for patients with relapsed disease > 100 days after completion of HDC)

  * Cytoreduction plus HDC is considered 1 chemotherapy regimen
* No other concurrent chemotherapy

Endocrine therapy

* At least 7 days since prior steroids

Radiotherapy

* More than 3 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior major surgery

Other

* Use of antibiotics for marginal zone lymphoma does not count as a prior therapy
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2002-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety
Efficacy

SECONDARY OUTCOMES:
Progression-free survival
Mean and median duration of response
Mean and median duration of progression-free and overall survival
Probability of polymerase chain reaction negativity after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Owen A. O'Connor, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont